March 26, 2019

Evaluation of Plasma Cholecystokinin (CCK) Levels and Gallbladder (GB) Functions in Hyperemesis Gravidarum

NCT 03950167.

#### INFORMED CONSENT FORM

We invite you to the research titled "Evaluation of Gallbladder Function and Cholecystokinin Level in Pregnant Women Diagnosed with Hyperemesis Gravidarum" conducted by Müge Keskin and Gamze Sinem Çağlar. Participation in this study is completely voluntary. You have the right not to participate in the study or to withdraw from the study at any time after participating. You will not be charged any fee for your participation in this study. The information to be obtained from this study will be used purely for research purposes and your personal information will be kept confidential.

# Aim of the study

Aim of the study is, evaluation of gallbladder functions and cholecystokinin hormone levels in patients with severe nausea and vomiting associated with pregnancy. You are taking part in the study as a participant of control group (healthy pregnant women )/ study group (pregnant women with nausea and vomiting of pregnancy) Your results will be compared to the study/control group. After fasting for 12 hours, you will be invited to hospital to get blood tests then you will be asked to eat 100 g milk chocolate (obtained by us), afterwards you will again donate blood sample for the analysis.

Your gallbladder will be evaluated by transabdominal ultrasound before and after eating chocolate.

#### Content of the Research

Your diagnosis and treatment will not be interfered with within the scope of the study.

If you do not want to participate in the study or if you want to leave the study, there will be no disruption or change in your treatment.

## **Reason for Research**

Scientific research

## **Expected Duration of the Research**

The duration of the study is 6 months and patient follow-up will not be required.

#### Places of Research

Ufuk University Faculty of Medicine Department of Obstetrics and Gynecology

## PARTICIPANT STATEMENT

It was stated that the research titled "Evaluation of Gallbladder Function and Cholecystokinin Level in Pregnant Women Diagnosed with Hyperemesis Gravidarum" will be conducted, and the above information about this research was conveyed. After this information, I was invited as a participant in the study. If I agreed to participate in this study, I was assured that my identity would be kept confidential both during the conduction and publication of the study. I consent to the use of my data. I have been given sufficient confidence that my personal information will be carefully protected during the use of research results for educational and scientific purposes. I can withdraw without giving any reason during the conduction of the research. I do not take any financial responsibility for the expenses to be made for the research. No payment will be made to me. I have fully understood all the explanations made to me regarding the research. I participate in this study with my own personal consent, without any pressure.

Name of the participant, date, signature